CLINICAL TRIAL: NCT04926922
Title: PREVAIL VIIIa: Evaluation of Latent Tuberculosis Infection Screening Methods in People Living With Retroviral Infection in Liberia
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000231; 000231-I
Record Dates: First submitted 2021-06-12; First posted 2021-06-15 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12-03

CONDITIONS: Tuberculosis; HIV
Keywords: Interferon-Gamma Release Assay (IGRA); Purified Protein Derivative (PPD); Tuberculin Skin Test (TST); TB; HIV; Natural History
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HONOR TB participants with positive IGRA and/or TST during initial phase: Adult participants who who tested positive on IGRA and or TST during initial phase and meet the study-specific eligibility criteria.

SUMMARY:
Background:

Tuberculosis (TB) is a health threat for people living with human immunodeficiency virus (HIV). People living with HIV are more likely than others to develop active TB. Also, TB makes HIV progress faster. TB is a leading cause of death among people in the West African country of Liberia. Researchers want to find an effective testing method for latent tuberculosis infection (LTBI) to help people living with HIV in Liberia.

Objective:

To compare the interferon-gamma release assay (IGRA) and tuberculin skin test (TST) as LTBI screening tests in people living with HIV in Liberia.

Eligibility:

People ages 18 and older who take part in NIH study #19-I-N014 and are scheduled to have or have had IGRA at a Month 12 HONOR study visit.

Design:

Participants will be screened with a medical history and physical exam. Their medical records and HONOR study records will be reviewed.

Participants will have TST. Purified protein derivative will be placed in the skin of their forearm. They will be observed for adverse reactions for 15 minutes. Between 48 and 72 hours after placement, they will have a second study visit to have the TST read. If they miss this time frame, they can return up to 7 days after placement. If they have a positive test result, they will have a chest x-ray. They will have a third study visit to review the results of the chest x-ray. They will be referred for clinical care if needed. They will take a pregnancy test if needed.

Participation will last from 2 days to 6 weeks.

DETAILED DESCRIPTION:
Study Description:

This is a prospective study to compare the interferon-gamma release assay (IGRA) and tuberculin skin test (TST) as latent tuberculosis infection (LTBI) screening tests in people living with HIV in Liberia. Participants will be co-enrolled on the ongoing HONOR (A CoHOrt Clinical, Viral, and ImmuNOlogic Monitoring Study of People Living with Retroviral Infection in Liberia) study. A TST will be administered to eligible participants who are being screened by IGRA on HONOR. Since there is no gold standard for diagnosing LTBI, the results of each method will be compared to evaluate whether there is no difference in the probability of testing positive, assess the operational functionality in the clinic and lab, and determine whether one test can be used with greater sensitivity assuming comparable specificity.

In an extension phase, participants who had a positive TST and/or IGRA result will be offered an opportunity to return for an optional assessment by follow-up chest x-ray, non-contrast chest computed tomography (CT) scanning, sputum collection, and phlebotomy. This will involve an additional visit (Visit 4), to occur after completion of the primary phase (Visit 3). The visit may occur in conjunction with (ie, the same day as or within 4 weeks of) a main HONOR study visit, and results of blood tests collected under the main HONOR study will be reviewed. For participants who have already completed the main HONOR study or do not have an upcoming HONOR visit scheduled, a new visit (ie, HONOR TB Visit 4) will be scheduled for this HONOR TB extension study, and a blood draw will also be performed.

Objectives:

Primary Objective: Assess the sensitivity of the IGRA and TST as LTBI screening tools in people living with HIV in Liberia.

Secondary Objective: Assess the operational functionality of the IGRA and TST in Liberia.

Exploratory Objective: Investigate testing approaches, including follow-up chest x-ray imaging, high-resolution chest CT imaging, and performance on sputum of the Mycobacterium tuberculosis (MTB) complex/rifampin (RIF) nucleic acid amplification test (NAAT), to improve diagnosis of stage-specific TB infection by examining how classification of TB status is associated with biomarker levels (only for participants with a positive TST and/or IGRA).

Endpoints:

Primary Endpoint: Frequency of positive results using the IGRA and TST.

Secondary Endpoint: Proportion of each test type successfully completed and the result determined.

Exploratory Endpoint: Repeat chest x-ray assessment, non-contrast chest CT assessment, sputum analysis by MTB/RIF NAAT assay, and analysis of serum by a CRISPR-Mtb-cfDNA assay.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Be a participant on the PREVAIL VIII/HONOR study.
* Be at least 18 years of age.
* Be scheduled to undergo or have undergone IGRA at a Month 12 HONOR study visit.
* Ability to return to the clinic 48 to 72 hours after TST placement for reading.
* Ability to provide informed consent.

In order to be eligible to participate in the extension phase of the study, an individual must meet all of the following criteria:

* Participated in the PREVAIL VIIIa HONOR TB study.
* Have had a positive TB test result on the TST and/or IGRA performed as part of the PREVAIL VIII HONOR or PREVAIL VIIIa HONOR TB study(ies).
* Ability to provide informed consent.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this

study:

* Received BCG vaccine <=10 years prior.
* Known hypersensitivity or allergy to any component of the PPD product.
* Previous severe reaction (e.g., necrosis, blistering, ulcerations, or anaphylactic shock) to a TST.
* Documented active TB or a clear history of treatment for latent infection or active disease.
* Extensive burns or eczema or other skin conditions on the forearms that could affect placement and reading of the TST.
* Pregnant or lactating women.
* Any condition that, in the opinion of the investigator, would compromise the safety of the study participant or staff, or would prevent proper conduct of the study.

An individual who meets any of the following criteria will be excluded from participation in the extension phase of this study:

* Pregnant women.
* Contraindication to CT scanning.
* Any condition that, in the opinion of the investigator, would compromise the safety of the study participant or staff, or would prevent proper conduct of the study.

Exclusion of Special Populations (Children, Adults Who Lack Capacity to Consent, and Pregnant Women)

-We are able to obtain knowledge about TST performance in Liberia without exposing children, adults who lack capacity to consent, and pregnant women to the potential risk of reactions to the TST or exposure to radiation for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants must be enrolled in the main HONOR study of people living with HIV in Liberia who participated in the HONOR TB study at their Month 12 visit and tested positive on IGRA and/or TST.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2026-06-07 (Estimated); Study Completion 2026-06-07 (Estimated)

PRIMARY OUTCOMES:
Frequency of positive results using the IGRA and TST. | 48-72 hours after TST placement
  Assess the sensitivity of the IGRA and TST as LTBI screening tools in people living with HIV in Liberia.

SECONDARY OUTCOMES:
Proportion of each test type successfully completed and the result determined. | 48-72 hours after TST placement
  Assess the operational functionality of the IGRA and TST.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Migueles, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (5):
- National Institutes of Health Cinical Center, Bethesda, Maryland, United States
- Liberia (4):
  - C.H. Rennie Hospital, Kakata
  - Duport Road Clinic, Monrovia
  - JFK Medical Center, Monrovia
  - Redemption Hospital, Monrovia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. Utilized for individual participant data meta-analysis. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our database but without investigator support.